CLINICAL TRIAL: NCT06707350
Title: Protective Effect of Remote Ischemic Preconditioning (RIPC) Against Negative Inflammatory Response and Organ Dysfunction After Cardiovascular Surgery (Panda VII)
Brief Title: Protective Effect of RIPC Against Negative Inflammatory Response and Organ Dysfunction After Cardiovascular Surgery (Panda VII)
Acronym: PANDA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of China 5A Network, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PANDA VII
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cardiopulmonary Bypass; Cardiovascular Diseases; Inflammatory Response During Cardiac Surgery
Keywords: inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIPC Group (Experimental): 6 cycles of 5-minute inflation and 5-minute deflation on 2 upper and lower libms with a blood pressure cuff at 72, 36, 24 hours before surgery
  Interventions: Device: Remote ischemic preconditioning (RIPC)
- Control group (Sham Comparator): 8 cycles of 5-minute inflation to a pressure of 20 mm Hg followed by 5-minute cuff deflation on 2 upper and lower libms with a blood pressure cuff at 72, 36, 24 hours before surgery
  Interventions: Device: sham condition (control group)

INTERVENTIONS:
Device: Remote ischemic preconditioning (RIPC) — 8 cycles of 5-minute inflation and 5-minute deflation on 2 upper and lower limbs with a blood pressure cuff
  Arms: RIPC Group
Device: sham condition (control group) — 8 cycles of 5-minute inflation to a pressure of 20 mm Hg followed by 5-minute cuff deflation.
  Arms: Control group

SUMMARY:
Remote ischaemic pre-conditioning (RIPC) has been recognized as a low-cost, non-invasive intervention method by applying brief ischaemia and reperfusion on an arm or a leg. Previous studies have mainly focused on the organoprotective effects of RIPC in patients undergoing cardiac surgery. However, whether it has an organ-protecting effect is still highly debated. We aimed to determine whether intensive RIPC can prevent from negative inflammatory response and organ dysfunction as well as postoperative complications in patients undergoing cardiovascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients at high risk for organ dysfunctions who underwent elective cardiovascular surgery requiring cardiopulmonary bypass (CPB);
* age of 18 -80 years old, regardless of gender;
* subjects voluntarily participate in the trialand sign the informed consent;

Exclusion Criteria:

* 1) Arm fracture, skin injury or infection;
* 2) There is limb nerve injury;
* 3) Limb placement PICC, arteriovenous fistula and other devices that affect armband placement;
* 4) There are basic vascular lesions and poor blood supply at the extremities;
* 5) Limb thrombosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
∆SOFA | within the prior 7 days after cardiac surgery.
  the change in sequential organ failure assessment score [∆SOFA]) was defined as the difference between the mean total postoperative SOFA score, calculated maximally to the 9th postoperative day, and the basal SOFA score.

SECONDARY OUTCOMES:
Plasma interleukin-1 levels | within the prior 7 days after cardiac surgery.
  Plasma interleukin-1 levels within the prior 7 days after cardiac surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-feng Shao, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jia P, Ji Q, Zou Z, Zeng Q, Ren T, Chen W, Yan Z, Shen D, Li Y, Peng F, Su Y, Xu J, Shen B, Luo Z, Wang C, Ding X. Effect of Delayed Remote Ischemic Preconditioning on Acute Kidney Injury and Outcomes in Patients Undergoing Cardiac Surgery: A Randomized Clinical Trial. Circulation. 2024 Oct 22;150(17):1366-1376. doi: 10.1161/CIRCULATIONAHA.124.071408. Epub 2024 Sep 25. PMID 39319450